CLINICAL TRIAL: NCT01000207
Title: A Multi-center, Randomized, Single-blind, Dose-Ranging Study to Evaluate Immunogenicity, Safety and Tolerability of Different Doses of Adjuvanted Cell-Derived, Inactivated Novel Swine Origin A/H1N1 Monovalent Subunit Influenza Virus Vaccine in Healthy Japanese Pediatric Subjects
Brief Title: Single-blind, Dose-ranging Study of Novel Swine Influenza Virus Vaccine in Japanese Pediatric Subjects
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V110_08
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2012-01

CONDITIONS: Swine-Origin Influenza A H1N1 Virus
Keywords: Influenza A; H1N1 subtype; Children/adolescent; Vaccine; Adjuvant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Dose ranging
  Interventions: Biological: Adjuvanted cell-derived, inactivated novel swine origin A/H1N1 monovalent subunit influenza virus vaccine
- 2 (Experimental): Dose ranging
  Interventions: Biological: Adjuvanted cell-derived, inactivated novel swine origin A/H1N1 monovalent subunit influenza virus vaccine

INTERVENTIONS:
Biological: Adjuvanted cell-derived, inactivated novel swine origin A/H1N1 monovalent subunit influenza virus vaccine — High dose group and low dose group of adjuvanted vaccines

SUMMARY:
This study is to identify the preferred vaccine dosage (of antigen and adjuvant) and schedule (one or two administrations) of the cell-derived H1N1sw monovalent vaccine in healthy children/adolescents based on European Medicines Agency's Committee for Medicinal Products for Human Use (EMEA/CHMP) criteria, and safety and tolerability.

DETAILED DESCRIPTION:
This is a multi-center, randomized, single-blind, dose-ranging study. Subjects were randomized at a 1:1 ratio to receive either 3.75μg of cell-derived H1N1sw vaccine formulated in half (i.e., half the content of the European-licensed adjuvanted seasonal influenza vaccine) MF59 adjuvant (3.75_halfMF59) or 7.5μg of cell-derived H1N1sw vaccine formulated with full MF59 (7.5_fullMF59). Subjects were not informed of their allocated doses. Two vaccinations were administered IM three weeks apart. Subjects in both the vaccine groups were stratified into three age strata: 6 to 35 months, 3 to 8 years and 9 to 19 years. Blood samples were collected at day 1 (baseline), three weeks after the first vaccination (day 22) and three weeks after the second vaccination (day 43). Sera were tested by Hemagglutination Inhibition (HI) and Microneutralization (MN) assays. Local and systemic reactions were collected for the first week following each injection using Diary Card (i.e., day 1 to day 7 and day 22 to day 28). All adverse events (AE), serious adverse events (SAE), and AEs that led to withdrawal from the study and related prescription medications were collected for the entire study period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese aged 6 months to 19 years

Exclusion Criteria:

* History of anaphylaxis, serious vaccine reactions, hypersensitivity to vaccine viral proteins or excipients
* Administration of adjuvanted influenza vaccine or suspected influenza disease within 3 month prior to study start
* Administration of any other vaccines within 4 weeks prior to enrollment expect for seasonal influenza vaccines within 1 week
* History of progressive or severe neurological disorders

Ages: 6 Months to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 123 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Seroprotection, GMRs and Seroconversion rate at Weeks 0, 3 and 6 | 6 weeks

SECONDARY OUTCOMES:
AEs, vital signs, laboratory tests | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- Sites 1,2,3,4,5, Kagoshima, Japan

REFERENCES:
- [Result] Yasuda Y, Komatsu R, Matsushita K, Minami T, Suehiro Y, Sawata H, Nakura N, Jaeger RK, Lattanzi M. Comparison of half and full doses of an MF59-adjuvanted cell culture-derived A/H1N1v vaccine in Japanese children. Adv Ther. 2010 Jul;27(7):444-57. doi: 10.1007/s12325-010-0043-4. Epub 2010 Jun 25. PMID 20586002